CLINICAL TRIAL: NCT04447872
Title: Prospective, Randomized Trial Comparing Luteal Phase Ovarian Stimulation, and Luteal Estradiol Priming Protocol for Patients With Diminished Ovarian Reserve - The LUTEAL Trial
Brief Title: The LUTEAL Trial: Luteal Stimulation vs. Estrogen Priming Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Mary Rausch, MD, Assistant Professor, Donald and Barbara Zucker School of Medicine at Hofstra/Northwell, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0080
Record Dates: First submitted 2020-06-18; First posted 2020-06-25 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Infertility; Diminished Ovarian Reserve; IVF
Keywords: IVF; In Vitro Fertilization; DOR; Diminished Ovarian Reserve; Controlled ovarian stimulation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luteal phase ovarian stimulation (LPOS) (Active Comparator): Patients will present in the luteal phase, and will begin 150 IU hMG and 300 IU recombinant FSH daily, as well as oral Clomiphene citrate 100mg daily for the first five days of the stimulation. FSH can then be titrated per patient response. Gonadotropin releasing hormone antagonist (Ganirelix, Organon; and cetrorelix, Serono) will be started per criteria. Once patients are ready for ovulation trigger, 5-10,000 units of human chorionic gonadotropin, +/- GnRH agonist (i.e Luprolide acetate 40 IU), will be administered. All metaphase II oocytes obtained by oocyte retrieval will be fertilized with intracytoplasmic sperm injection (ICSI) or IVF. Embryos will be cultured to the blastocyst stage and vitrified on day 5-7 with or without embryo biopsy for genetic analysis.
  Interventions: Procedure: Timing of injectable gonadotropins
- Luteal estradiol priming protocol (Active Comparator): In the luteal phase, the patient will begin Estradiol patches 0.1mg QOD. She will also take daily Gonadotropin releasing hormone (GnRH) antagonist (Ganirelix, Organon; and cetrorelix, Serono) for three days. With menses, she will begin 150 IU hMG, 300 IU recombinant FSH daily, and oral Clomiphene citrate 100mg qd (for five days). FSH can be titrated per patient response. GnRH antagonist will be started per criteria. 5-10,000 units of human chorionic gonadotropin, +/- GnRH agonist (i.e Luprolide acetate 40 IU) will be administered for ovulation trigger. All metaphase II oocytes obtained by oocyte retrieval will be fertilized with intracytoplasmic sperm injection (ICSI) or IVF. Embryos will be cultured to the blastocyst stage and vitrified on day 5-7 with or without embryo biopsy for genetic analysis.
  Interventions: Procedure: Timing of injectable gonadotropins

INTERVENTIONS:
Procedure: Timing of injectable gonadotropins — Gonadotropins will with be started in the luteal phase or in follicular phase (preceded by Estradiol patches)

SUMMARY:
Ovarian reserve defines the quantity and quality of the ovarian primordial follicular pool. Diminished ovarian reserve (DOR) indicates a reduction in the quantity of ovarian follicular pool to less than expected for age. It is an important cause of infertility in many couples.

To date, there is no clear consensus in the literature on the definition of diminished ovarian reserve, and it is unclear whether low oocyte yield results from an abnormal atresia rate of the follicle pool, or from a lower follicle pool at birth or whether it can just occur as a normal variation in the population.

The ovarian response to controlled ovarian stimulation with gonadotropins (for example, for in vitro fertilization) is largely determined by the ovarian reserve, and there are numerous different ovarian stimulation protocols that are employed to try and increase the oocyte yield of a particular cycle. There is no consensus on which, if any, of these protocols are superior and preferred for patient with DOR.

Luteal gonadotropin stimulation is a protocol of controlled ovarian stimulation (COS) for use in assisted reproductive technologies (ART) that has emerged over the past decade as an acceptable alternative to the classic follicular gonadotropin stimulation.

The luteal estradiol patch protocol was introduced in 2005 in patients with poor response to controlled ovarian stimulation (COS) and to address the phenomenon of early follicle recruitment in patients with diminished ovarian reserve (DOR). Luteal gonadotropin stimulation can potentially achieve the same effect by initiating follicular recruitment for IVF prior to the body's own premature recruitment.

Our hypothesis is that the luteal stimulation protocol and estradiol priming protocol are equivalent with regard to the outcome of number of mature oocytes retrieved. Patients who will be undergoing controlled ovarian stimulation and who have a diagnosis of diminished ovarian reserve will be considered for this trial, and enrolled if meeting all inclusion and no exclusion criteria.

DETAILED DESCRIPTION:
Patients who will be undergoing controlled ovarian stimulation and who have a diagnosis of diminished ovarian reserve will be considered for this trial, and enrolled if meeting all inclusion and no exclusion criteria. Patients will be randomized to one of two possible stimulation cycles as will be described.

Luteal Phase Ovarian Stimulation (LPOS)

Patients will present for an appointment on approximately day 15-18 of her menstrual cycle. If serum progesterone >3 ng/mL, and bHCG < 5 mIU/mL, the patient will begin 450 IU of daily injectable gonadotropins: 150 IU of hMG (Menopur®, Ferring Pharmaceuticals) and 300 IU of recombinant FSH (rFSH) (Gonal F®,Serono; or Follitropin beta (Follistim®, Organo)). The specific rFSH chosen will be based on the individual patient's insurance coverage. The patient will perform daily injections during the course of her stimulation, and will also take oral Clomiphene citrate 100mg daily for the first five days of the stimulation. FSH dose will be titrated during the stimulation (per physician discretion) based on serum estradiol levels and ovarian response to a minimum of no gonadotropins and a maximum of 600 IU daily. She will present for follicular monitoring ultrasound and serum blood tests on stimulation day 3-4, 5-6, and 7-8-~15. Gonadotropin releasing hormone (GnRH) antagonist (Ganirelix, Organon; and cetrorelix, Serono) will be started daily once either (1) serum estradiol level reaches > 400 pg/mL, lead follicle size > 13mm, or (2) on stimulation day 6. Once patient are ready for ovulation trigger as determine by physician, 5-10,000 units of human chorionic gonadotropin (Novarel®: Ferring Pharmaceuticals; or Pregnyl®: Schering-Plough) will be administered. A patient's trigger shot could be changed to include a GnRH agonist (i.e Luprolide acetate 40 IU) if deemed clinically necessary for ovarian hyperstimulation syndrome prevention. On the morning after hCG administration, patients' blood will be drawn and serum analyzed for hCG concentration to ensure adequate absorption (mean time 8-10 hours). Transvaginal oocyte retrieval will be performed 35 to 37 hours after hCG trigger. All metaphase II oocytes will be fertilized with intracytoplasmic sperm injection (ICSI) or IVF per patient request and laboratory protocol. Embryos will be cultured to the blastocyst stage and vitrified on day 5-7. If patient requests preimplantation genetic testing for aneuploidy (PGT-A), an embryo biopsy will be performed on day 5-7 of development prior to vitrification, and biopsy specimen will be sent to an outside laboratory for chromosome analysis.

Luteal Estradiol priming protocol (E2 prime)

Patients will present for an appointment on approximately day 18-21 of her menstrual cycle. If serum progesterone >3 ng/mL, and bHCG < 5 mIU/mL, the patient will begin Estradiol patches (Vivelle Dot 0.1mg, Novartis Pharmaceuticals; or Climara, Bayer) and change them every other day. She will also take daily Gonadotropin releasing hormone (GnRH) antagonist (Ganirelix, Organon; and cetrorelix, Serono) for the following three days.

Patients will then present for a baseline appointment with onset of her menses. If serum progesterone < 1.0 ng/mL, and bHCG < 5 mIU/mL, on cycle day 2-3 the patient will stop her estrogen patches and start 450 IU of daily injectable gonadotropins: 150 IU of hMG (Menopur®, Ferring Pharmaceuticals) and 300 IU of recombinant FSH (rFSH) (Gonal F®,Serono; or Follitropin beta (Follistim®, Organo)). The specific rFSH chosen will be based on the individual patient's insurance coverage. Estrogen patch will be removed the day of starting gonadotropin injections. The patient will perform daily injections during the course of her stimulation, and will also take oral Clomiphene citrate 100mg daily for the first five days of the stimulation. FSH dose will be titrated during the stimulation (per physician discretion) based on serum estradiol levels and ovarian response to a minimum of no gonadotropins and a maximum of 600 IU daily. She will present for follicular monitoring ultrasound and serum blood tests on stimulation day 3-4, 5-6, and 7-8-~15. Gonadotropin releasing hormone (GnRH) antagonist (Ganirelix, Organon; and cetrorelix, Serono) will be started daily once either (1) serum estradiol level reaches > 400 pg/mL, lead follicle size > 13mm, or (2) on stimulation day 6. Once patient are ready for ovulation trigger as determine by physician, 5-10,000 units of human chorionic gonadotropin (Novarel®: Ferring Pharmaceuticals; or Pregnyl®: Schering-Plough) will be administered. A patient's trigger shot could be changed to include a GnRH agonist (i.e Luprolide acetate 40 IU) if deemed clinically necessary for ovarian hyperstimulation syndrome prevention. On the morning after hCG administration, patients' blood will be drawn and serum analyzed for hCG concentration to ensure adequate absorption (mean time 8-10 hours). Transvaginal oocyte retrieval will be performed 35 to 37 hours after hCG trigger. All metaphase II oocytes will be fertilized with intracytoplasmic sperm injection (ICSI) or IVF per patient request and laboratory protocol. Embryos will be cultured to the blastocyst stage and vitrified on day 5-7. If patient requests preimplantation genetic testing for aneuploidy (PGT-A), an embryo biopsy will be performed on day 5-7 of development prior to vitrification, and biopsy specimen will be sent to an outside laboratory for chromosomal analysis.

Outcomes between the two stimulation protocols will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Female aged 20 - 45
4. Regular menstrual cycles between 21 and 40 days
5. Presence of both ovaries
6. Meets criteria for DOR by the recent ASRM/ACOG Committee Opinion

   1. antimüllerian hormone (AMH) value less than 1 ng/mL
   2. antral follicle count less than 5-7 and
   3. follicle-stimulating hormone (FSH) greater than 10 IU/L or
   4. a history of poor response to in vitro fertilization stimulation (fewer than four oocytes at time of egg retrieval).

Exclusion Criteria:

1. Oocyte donation cycle
2. Oocyte freezing cycle
3. Current ovarian cyst > 3cm
4. Anovulatory or oligo-ovulatory (<6 ovulation per year)
5. Previous oophorectomy
6. Exposure to cytotoxic or pelvic irradiation
7. Planned aromatase inhibitor usage during current ovarian stimulation
8. Sensitizing or ovarian stimulating therapy in the past one month

   Additional contraindications to this study re, as follows (because such patients cannot receive an estrogen patch):
9. Undiagnosed abnormal genital bleeding
10. Known, suspected, or history of breast cancer
11. Known or suspected estrogen-dependent neoplasia
12. Active DVT, PE, or a history of these conditions
13. Active arterial thromboembolic disease (for example, stroke and MI), or a history of these conditions
14. Known anaphylactic reaction or angioedema with estradiol patches
15. Known liver impairment or disease
16. Known protein C, protein S, or antithrombin deficiency, or other known thrombophilic disorders

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of mature (Metaphase II) oocytes retrieved | First day after oocyte retrieval
  Mature oocytes, capable of being fertilized in vitro

SECONDARY OUTCOMES:
Number of oocytes cumulus complexes retrieved | First day after oocyte retrieval
  Total oocytes from oocyte retrieval
Oocyte fertilization rate | First day after oocyte retrieval
  Rate of oocytes that develop two pronuclei
Blastocyst development rate | Day 5-7 following oocyte retrieval
  Rate of embryos that develop to the blastocyst stage
Cycle cancellation rate | Within two weeks of cycle start
  Rate of cycle cancellation prior to oocyte retrieval
Total FSH dosage (IU) used | From the first day of injections, through the day of oocyte retrieval
  Total dosage of injected gonadotropins during ovarian stimulation
Duration of stimulation (days) | From the first day of injections, through the day of oocyte retrieval
  How many days from first injection until trigger shot injection

OTHER OUTCOMES:
Embryo ploidy status | When biopsy results return, usually within four weeks after oocyte retrieval
  If patient undergoes preimplantation for genetic testing of aneuploidy (PGT-A), we will compare the rate of euploid embryos between the groups
Implantation rate | Two weeks post embryo transfer
  Rate of successful embryo implantation if undergoes embryo transfer
Clinical pregnancy rate | Five to seven weeks post embryo transfer
  Rate of successful clinical intrauterine pregnancy if undergoes embryo transfer
Live birth rate | 40 weeks post embryo transfer
  Rate of live birth if undergoes embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Fertility, Manhasset, New York, United States

REFERENCES:
- [Background] Lin LT, Vitale SG, Chen SN, Wen ZH, Tsai HW, Chern CU, Tsui KH. Luteal Phase Ovarian Stimulation May Improve Oocyte Retrieval and Oocyte Quality in Poor Ovarian Responders Undergoing In Vitro Fertilization: Preliminary Results from a Single-Center Prospective Pilot Study. Adv Ther. 2018 Jun;35(6):847-856. doi: 10.1007/s12325-018-0713-1. Epub 2018 Jun 4. PMID 29869107
- [Background] Zhang W, Wang M, Wang S, Bao H, Qu Q, Zhang N, Hao C. Luteal phase ovarian stimulation for poor ovarian responders. JBRA Assist Reprod. 2018 Sep 1;22(3):193-198. doi: 10.5935/1518-0557.20180045. PMID 29931967
- [Background] Wei LH, Ma WH, Tang N, Wei JH. Luteal-phase ovarian stimulation is a feasible method for poor ovarian responders undergoing in vitro fertilization/intracytoplasmic sperm injection-embryo transfer treatment compared to a GnRH antagonist protocol: A retrospective study. Taiwan J Obstet Gynecol. 2016 Feb;55(1):50-4. doi: 10.1016/j.tjog.2015.07.001. PMID 26927248
- [Background] Wu Y, Zhao FC, Sun Y, Liu PS. Luteal-phase protocol in poor ovarian response: a comparative study with an antagonist protocol. J Int Med Res. 2017 Dec;45(6):1731-1738. doi: 10.1177/0300060516669898. Epub 2017 Jan 16. PMID 28661216